CLINICAL TRIAL: NCT01619631
Title: Tai Chi Intervention for Chinese Americans With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Albert Yeung, Research Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011P001313; R21AT006123-01A1 (NIH)
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Depression
Keywords: Depression; Tai Chi; Alternative medicine; Mind body medicine
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 12-week Tai Chi intervention (Experimental)
  Interventions: Behavioral: 12-week Tai Chi intervention
- Education control group (Active Comparator): After 24 weeks, and upon completion of the study, each participant will be offered twelve weeks of Tai Chi twice weekly.
  Interventions: Behavioral: Education control group
- Waitlist control group (No Intervention): The waitlist control will not receive any intervention during the duration of the study. After 24 weeks, and upon completion of the study, each participant will be offered twelve weeks of Tai Chi twice weekly.

INTERVENTIONS:
Behavioral: 12-week Tai Chi intervention — Tai Chi classes will be conducted weekly for one hour each for 12 weeks. Classes will begin with warm-up exercises designed to loosen the body, increase awareness of alignment and structural integration, improve efficiency of breathing, incorporate mindfulness and imagery into movement.
  Arms: 12-week Tai Chi intervention
Behavioral: Education control group — The education control group will meet twice weekly for 12 weeks for one hour, and research staff will present didactic information modified from psychoeducation curriculums created by the Benson Henry Institute and a stress reduction study for depressed minority patients.
  Arms: Education control group

SUMMARY:
The purpose of this study is to conduct a pilot randomized controlled trial (RCT) that provides the feasibility, safety, and preliminary efficacy data required to design a large scale trial evaluating Tai Chi for Chinese Americans with major depressive disorder (MDD) who are not on antidepressant medications.

DETAILED DESCRIPTION:
Aim #1: To evaluate the feasibility and safety of conducting a RCT of Tai Chi for Chinese American adults with MDD who are not on antidepressant medications. The investigators hypothesize that: a) the investigators can develop a Tai Chi intervention and depression-related measurement protocol for Chinese Americans with MDD; b) the investigators will be able to recruit non-pharmacologically treated Chinese Americans with MDD to participate in a randomized controlled Tai Chi study; c) participants will be compliant with the Tai Chi intervention and all testing protocols; d) the Tai Chi intervention will be safe and study staff will be able to effectively monitor participants' depressive symptoms and assure their safety during the study.

Aim #2: To collect preliminary data on the efficacy of a 12-week Tai Chi group intervention for Chinese Americans with MDD who are not on antidepressant medications to determine the effect size needed for a definitive RCT. The investigators hypothesize that at the conclusion of 12-weeks, Tai Chi participants, as compared to control subjects, will demonstrate a) greater improvement in depressive symptoms (Hamilton Depression Severity Index-17, Beck Depression Inventory), b) greater improvement in functional status, general health, and well being (Clinical Global Impressions Scale, The SF-36 Health Survey (SF-36®) for social functioning, Exercise Self-Efficacy, Mindfulness), and c) greater social support (Multidimensional Scale of Perceived Social Support).

Aim #3: To characterize participants' experience in a trial of Tai Chi for Chinese Americans with MDD in order to optimally design a subsequent, more definitive study. Using mixed methods (qualitative and quantitative analyses), the investigators will identify the ethnocultural experience of Tai Chi among Chinese Americans with MDD, assess whether they view Tai Chi a more culturally acceptable alternative to conventional antidepressant therapy, explore the facilitators and barriers to adherence to the Tai Chi training protocol, identify characteristics of responders and non-responders to the Tai Chi intervention, and assess participants' willingness/intention to continue practice of Tai Chi beyond the study period. The investigators hypothesize that a) characteristics such as severity of illness, age, co-morbidities, and education level may distinguish responders from non-responders; b) participants with greater levels of class attendance and home practice will exhibit greater improvements in depressive symptoms; and c) participants who continue to practice Tai Chi after the 12-week training will maintain clinical improvements in depressive symptoms and a lower rate of relapse at the end of 3 additional months of follow-up compared to those who do not continue Tai Chi practice.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as being of Chinese ethnicity and fluent in Mandarin and/or Cantonese
* 18-80 years of age
* Satisfy DSM-IV criteria for MDD
* Baseline score of 14-20 on the 17-item Hamilton Rating Scale for Depression (HAM-D-17)
* No regular (≥ 3 times/week for ≥ 2 months) Tai Chi training/practice or other forms of mind-body intervention in the past 6 months

Exclusion Criteria:

* Primary psychiatric diagnosis other than MDD
* History of psychosis, mania, or severe cluster B personality disorder, active ETOH or substance abuse/dependency disorder in the past 6 months
* Unstable medical conditions as judged by investigators
* Use or plan to use confounding treatments, including antidepressants and CAM treatments thought to have beneficial effects on mood, such as St. John's Wort, S-Adenosyl methionine (SAMe), omega-3 fatty acids, light therapy, conventional psychotherapy, mind-body interventions (e.g. Qigong, mindfulness training, muscle relaxation training, etc.)
* Current active suicidal or self-injurious potential necessitating immediate treatment
* Women who are pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Major depressive disorder response rate, as determined by Hamilton Rating Scale for Depression (HAM-D 17-item) | Baseline, 12-weeks, 24-weeks
  Response will be defined as having a 50% or greater improvement in HAM-D-17 score at the conclusion fo treatment, compared to baseline.
Major depressive disorder remission as measured by DSM-IV and Hamilton Rating Scale for Depression (HAM-D 17-item) | Week 12, week 24
  Remission will require jointly the absence of the core symptoms of depression, with neither of the core features of DSM-IV depression (depressed mood or anhedonia) being reported at the threshold or subthershold level (using Chinese Bilingual SCID I/P interview) and HAM-D-17 score <8.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yeung, MD, ScD, Principal Investigator — Massachusetts General Hospital Depression Clinical and Research Program
Locations (2):
- United States (2):
  - South Cove Community Health Center, Boston, Massachusetts
  - Massachusetts General Hospital Depression Clinical and Research Program, Boston, Massachusetts

REFERENCES:
- [Background] Short KH, Johnston C. Stress, maternal distress, and children's adjustment following immigration: the buffering role of social support. J Consult Clin Psychol. 1997 Jun;65(3):494-503. doi: 10.1037//0022-006x.65.3.494. PMID 9170773
- [Background] Taylor-Piliae RE, Froelicher ES. Measurement properties of Tai Chi exercise self-efficacy among ethnic Chinese with coronary heart disease risk factors: a pilot study. Eur J Cardiovasc Nurs. 2004 Dec;3(4):287-94. doi: 10.1016/j.ejcnurse.2004.09.001. PMID 15572017
- [Background] Zhang J, Norvilitis JM. Measuring Chinese psychological well-being with Western developed instruments. J Pers Assess. 2002 Dec;79(3):492-511. doi: 10.1207/S15327752JPA7903_06. PMID 12511017
- [Derived] Yeung AS, Feng R, Kim DJH, Wayne PM, Yeh GY, Baer L, Lee OE, Denninger JW, Benson H, Fricchione GL, Alpert J, Fava M. A Pilot, Randomized Controlled Study of Tai Chi With Passive and Active Controls in the Treatment of Depressed Chinese Americans. J Clin Psychiatry. 2017 May;78(5):e522-e528. doi: 10.4088/JCP.16m10772. PMID 28570792